CLINICAL TRIAL: NCT02615327
Title: Verifying Fibers Meet Regulatory Definitions for Nutrition Facts Labeling: A Randomized, Controlled Trial Evaluating Polydextrose
Brief Title: Effect of Fiber on Glycemic Index
Acronym: Fiber2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB2015-104
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Fiber; Polydextrose; Glycemic Index
MeSH Terms: interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active Treatment 1 (Experimental): 8g Polydextrose
  Interventions: Dietary Supplement: 8 g Polydextrose
- Active Treatment 2 (Experimental): 12 g Polydextrose
  Interventions: Dietary Supplement: 12 g Polydextrose
- Active Treatment 3 (Experimental): 16 g Polydextrose
  Interventions: Dietary Supplement: 16 g Polydextrose
- Placebo (Placebo Comparator): 0 g Polydextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 8 g Polydextrose — 8g of Polydextrose
  Arms: Active Treatment 1
Dietary Supplement: 12 g Polydextrose — 12 g of Polydextrose
  Arms: Active Treatment 2
Dietary Supplement: 16 g Polydextrose — 16 g of Polydextrose
  Arms: Active Treatment 3
Dietary Supplement: Placebo — 0 g of Polydextrose
  Arms: Placebo

SUMMARY:
Primary objective is to investigate the effect of polydextrose on postprandial glucose concentrations in healthy adults when added to a food product.

Secondary objective is to assess gastrointestinal tolerance and acute bowel changes.

DETAILED DESCRIPTION:
This study is a randomized, 4-arm, single-blinded, controlled, cross-over trial design focused on determining the health benefits associated with Polydextrose intake.

A planned sample size of 40 will be enrolled into the study. This study will require one initial screening visit and 4 weekly study visits. This study will take approximately 4 weeks per subject to complete.

The initial screening visit will provide subject with the informed consent document and determine subject eligibility through anthropometric measurements, vital signs, fasting blood glucose test (finger prick), and completion of a survey relate to general eating, health, and exercise habits.

If willing and eligible to participate, subjects will be invited to participate in the study for 4 study days. Subjects will be instructed to maintain their usual diet pattern and physical activity throughout study duration. A dinner meal will be provided the day before the study visit to control the second meal effect from the food and beverage intake of the night before the study visit.

Subject will arrive at the center in a fasted state for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a Licensed health Care Professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Subjects will be randomized to receive a placebo or treatment beverage based on randomized treatment sequences for 4 study visits. The sequences of receiving the beverage treatments at each visit will be randomly assigned to one of sequences.

Each study visit will involve with blood samples collection at time points 0 (fasting), 0.5, 1, 2, 3 hour (h) for assessment of change in plasma glucose and insulin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged between 20 and 55 years of age
* Subject has BMI between 20.0 and 32.0 kg/m2 at screening visit
* Fasting blood sugar less than 126 mg/dL
* Subject is willing to maintain a stable body weight and to follow his/her regular diet and physical activity patterns throughout the study period.
* Subject is willing to refrain from vigorous physical activity and consumption of alcoholic and/or caffeinated beverages 24 h prior to each test day
* Subject does not smoke or has abstained from smoking for at least 2 years
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications or dietary supplements that would interfere with outcomes of the study.
* Subject typically consumes a low fiber diet that correlates with the average fiber intake of typical western diet.

Exclusion Criteria:

* Subject currently smokes or has smoked within the past 2 years
* Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compounds
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women with a fasting blood glucose concentration ≥126 mg/dL
* Average blood pressure > 140 mmHg/90 mmHg during screening visit
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years
* Men and women who are taking medication or dietary supplements that may interfere with the outcomes of the study. Subjects may choose to go off dietary supplements (requires 30 days washout)
* Men and women who have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months
* Substance (alcohol or drug) abuse within the last 2 years
* Excessive coffee and tea consumption (> 4 cups/day)
* Unstable weight: gained or lost weight +/- 5 lbs in previous 3 months
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study and women who are lactating.
* Men and women whom investigator is uncertain about subject's capability or willingness to comply with protocol requirements
* Special or atypical diet - eg. vegan, gluten free, excessively high or low energy/fiber
* Women who are taking unstable dose and brand of hormonal contraceptives and/or stable dose and brand less than 6 months.
* Men and women who do excessive exercise regularly or athlete

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-02-22 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Changes in plasma glucose concentration over a 3 hour Oral Glucose Tolerance Test (OGTT) after administration of polydextrose (8 g, 12g, 16 g) compared to 0 mg placebo | 3 hours
  3-hour Acute Postprandial plasma glucose Responses

SECONDARY OUTCOMES:
Changes in gastrointestinal tolerance using the questionnaire in 3 days following treatment administrations. | 3 days
  3 days after administration of each treatment
Changes in bowel movement using the questionnaire in 3 days following treatment administrations. | 3 days
  3 days after administration of each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Britt Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States